CLINICAL TRIAL: NCT04322760
Title: Effect of Lidocaine 5% Patch Supplementation to Intra-articular Bupivacaine Dexmedetomidine After Arthroscopic Knee Surgery Under General Anesthesia
Brief Title: Lidocaine 5% Patch Supplementation to Intra-articular Bupivacaine Dexmedetomidine After Arthroscopic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Said Elgebaly,MD, Assistant professor of Anesthesiology, Surgical Intensive Care, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31084/07/16
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Dexmedetomidine; Lidocaine 5% Patch; Arthroscopic Knee Surgery; Intra-articular
MeSH Terms: interventions — Lidocaine; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Patients were allocated into 2 groups, 20 patients in each received 10 ml 0.5 % bupivacaine and 1µg/kg dexmedetomidine diluted in 10 ml saline injected intra-articularly; group A: no patch, group B: a patch of lidocaine 5% was applied to the skin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control group) (Active Comparator): Patients in each received 10 ml 0.5 % bupivacaine and 1µg/kg dexmedetomidine diluted in 10 ml saline injected intra-articularly without lidocaine patch
  Interventions: Drug: Dexmedetomidine Bupivacaine
- Group B (Experimental): Patients in each received 10 ml 0.5 % bupivacaine and 1µg/kg dexmedetomidine diluted in 10 ml saline injected intra-articularly with a patch of lidocaine 5% was applied to the skin
  Interventions: Drug: Lidocaine 5% patch with Dexmedetomidine Bupivacaine

INTERVENTIONS:
Drug: Lidocaine 5% patch with Dexmedetomidine Bupivacaine — 10 ml 0.5 % Bupivacaine and 1µg/kg Dexmedetomidine diluted in 10 ml saline was injected intra-articularly through one of the arthroscopic ports after the end of the surgery under complete aseptic technique and a patch of lidocaine 5% was applied to the skin between the arthroscopic ports
  Arms: Group B
Drug: Dexmedetomidine Bupivacaine — 10 ml 0.5 % Bupivacaine and 1µg/kg Dexmedetomidine diluted in 10 ml saline was injected intra-articularly through one of the arthroscopic ports after the end of the surgery under complete aseptic technique without a patch of lidocaine 5%
  Arms: Group A (control group)

SUMMARY:
Surgery of the knee is a very common procedure which can be very painful and sufficient postoperative pain treatment is often problematic. The aim of this work was to study the effects of supplementation of intra-articular bupivacaine dexmedetomidine with lidocaine 5% patch after arthroscopic knee surgery under general anesthesia and its role in improving quality of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* ASA I & II
* Aged between 18 to 60 years
* Weight between 60 to 100 kg
* Scheduled for elective arthroscopic knee surgery

Exclusion Criteria:

* patient refusal.
* history of cardiac disease.
* impaired renal or hepatic function.
* hypertension treated with α methyldopa, clonidine, or beta-adrenergic blockers.
* if they have used opioid analgesics within the previous 24 hr.
* previous sensitivity to local anesthetics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The total dose of postoperative pethidine consumption | 24 hours
  The total dose of postoperative pethidine consumption; Pethidine 20 mg was given as rescue analgesia if pain visual analogue visual analogue scale (VAS) ≥4.

SECONDARY OUTCOMES:
First postoperative analgesia request time | 24 hours
  First postoperative analgesia (Pethidine 20 mg) request time
Pain intensity | 24 hours
  Visual analogue scale (VAS) was recorded immediately postoperative and at 30 min, 1, 2, 4, 6, 12 and 24 hours postoperatively. The score ranges from 0 to 10; higher means worse pain